CLINICAL TRIAL: NCT03343639
Title: A Randomized, Double-Blind, Placebo-Controlled Study of the Efficacy, Safety, and Tolerability of Serlopitant for the Treatment of Pruritus in Adults With Plaque Psoriasis
Brief Title: Study of the Efficacy, Safety and Tolerability of Serlopitant for the Treatment of Pruritus (Itch) With Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vyne Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MTI-109
Record Dates: First submitted 2017-11-10; First posted 2017-11-17 (Actual); Results first posted 2019-06-12 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Pruritus; Psoriasis
MeSH Terms: conditions — Pruritus; Psoriasis | interventions — serlopitant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 5 mg Serlopitant Tablets (Experimental): Serlopitant Tablets
  Interventions: Drug: 5 mg Serlopitant Tablets
- Matching Placebo Tablets (Placebo Comparator): Placebo Tablets
  Interventions: Drug: Matching Placebo Tablets

INTERVENTIONS:
Drug: 5 mg Serlopitant Tablets — Serlopitant Tablets
  Other Names: VPD-737
  Arms: 5 mg Serlopitant Tablets
Drug: Matching Placebo Tablets — Placebo Tablets
  Arms: Matching Placebo Tablets

SUMMARY:
Study of the efficacy, safety, and tolerability of serlopitant for the treatment of pruritus in adults with plaque psoriasis

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age 18-80 years at consent.
2. Diagnosis of plaque psoriasis for at least 6 months prior to randomization.

   a. Presence of plaque psoriasis in any anatomic location, covering ≤ 10% BSA in total, at the Screening and Baseline visits.
3. Pruritus of at least 4 weeks' duration prior to the initial Screening visit, and throughout the screening period prior to randomization.
4. Subjects must be willing to discontinue use of all psoriasis therapies other than the following, for the duration of the study: bland emollients (e.g., Cetaphil, Eucerin, Aquaphor) on any anatomic location; coal tar shampoos, limited to use on scalp.
5. WI-NRS initial screening score consistent with severe pruritus.
6. WI-NRS scores during the 2 weeks of screening consistent with sever pruritus.
7. All female subjects who are of childbearing potential must be willing to practice highly effective contraception (i.e., pregnancy prevention method with a failure rate of < 1% per year) from the time of the initial Screening visit until 2 weeks after last dose of study drug.
8. Weight ≥ 32 kg at the Screening and Baseline visits.
9. Willing and able to complete daily eDiary entries within a consistent timeframe for the duration of the study.

   1. Subjects must have ≥ 80% eDiary completion rate during the two weeks of the screening period immediately prior to randomization.

Exclusion Criteria:

1. Prior treatment with serlopitant.

   a. Prior treatment with other neurokinin-1 receptor (NK1-R) antagonists (e.g., aprepitant, fosaprepitant, rolapitant) is not allowed within 1 year prior to randomization.
2. Clinical worsening of psoriasis in the opinion of the investigator (e.g., increase in affected BSA or severity requiring use of systemic psoriasis therapies) within 12 weeks prior to randomization.
3. Predominance of non-plaque forms of psoriasis (e.g., guttate, drug-induced, pustular, erythrodermic).
4. Presence of any concurrent medical condition that provides a clearly defined etiology for pruritus other than psoriasis. These include but are not limited to urticaria, atopic dermatitis or other dermatologic conditions, hepatic or renal disease, psychogenic pruritus, drug reaction, untreated hyperthyroidism, and infection.
5. Treatment with systemic biologic therapies including but not limited to etanercept, infliximab, adalimumab, ustekinumab, secukinumab, or ixekizumab, within 6 months or 5 half-lives (whichever is longer) prior to randomization.
6. Treatment with systemic non-biologic psoriasis therapies, including but not limited to systemic corticosteroids, phosphodiesterase-4 inhibitors, Janus kinase inhibitors, cyclosporine, methotrexate, retinoids, hydroxyurea, mycophenolate mofetil, thioguanine, sirolimus, azathioprine, or fumaric acid derivatives, within 12 weeks prior to randomization.
7. Treatment with any of the following therapies within 4 weeks prior to randomization:

   a. Any topical/local psoriasis therapies other than those permitted per inclusion #4, including but not limited to topical corticosteroids, vitamin D analogues, calcineurin inhibitors, phosphodiesterase-4 inhibitors, Janus kinase inhibitors, non-shampoo forms of coal tar, salicylates, retinoids, anthralin, or excimer laser.

   i. Non-systemic corticosteroids that do not involve skin application (e.g., inhaled, intranasal, or intra-articular corticosteroids) will be permitted.

   b. Phototherapy, with or without psoralen. c. Use of an indoor tanning facility, or sun exposure likely to result in sunburn.

   d. Systemic therapies with recognized anti-pruritic properties including but not limited to H1 antihistamines, doxepin, mirtazapine, gabapentin, pregabalin, cannabinoids, and kappa opioid receptor agonists.

   e. Any topical anti-pruritic therapies, including but not limited to H1 antihistamines, doxepin, capsaicin, or medicated emollients (e.g., menthol or pramoxine).

   f. Strong CYP3A4 inhibitors.
8. Treatment with any investigational therapy within 4 weeks or 5 half-lives (whichever is longer) prior to randomization.
9. Serum creatinine, total bilirubin, alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2x the upper limit of normal (ULN) during screening.
10. History of malignancy within 5 years prior to randomization, with the exception of completely treated and non-metastatic basal cell carcinoma or squamous cell carcinoma of the skin.
11. Presence of any of the following conditions meeting DSM-5 diagnostic criteria within 3 years prior to randomization: major depressive disorder, bipolar disorder, schizophrenia, psychotic disorder, intellectual disability, severe alcohol use disorder, or other known psychiatric condition meeting DSM-5 diagnostic criteria which may confound the assessment of serlopitant safety or efficacy, compromise the safety of the subject, or interfere with the subject's ability to comply with protocol-mandated activities.
12. Suicidal ideation within 3 years prior to randomization, or history of suicide attempt at any time.
13. Known active hepatitis infection.
14. Known history of human immunodeficiency virus (HIV) infection.
15. Documented history of parasitic infection, including skin parasites such as scabies, within 12 months prior to randomization.
16. History of hypersensitivity to serlopitant or any of its components.
17. Currently pregnant or breastfeeding female subject.
18. Presence of any medical condition or disability that, in the investigator's opinion, could interfere with the assessment of serlopitant safety or efficacy, compromise the safety of the subject, or interfere with the subject's ability to comply with protocol-mandated activities; this includes any clinically significant screening ECG abnormalities any may include some clinically significant screening laboratory abnormalities.

    a. Unless specifically excluded per exclusion #9, clinically significant laboratory abnormalities at screening which are unlikely to interfere with the assessment of safety or efficacy in this trial, compromise the safety of the subject, or interfere with the subject's ability to comply with protocol mandated activities are permitted.
19. Planned or anticipated major surgical procedure or other activity that would interfere with the subject's ability to comply with protocol-mandated assessments (e.g., extended international travel) during the subject's participation in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-10-23 (Actual); Study Completion 2018-11-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (39):
- United States (39):
  - Study Site 221, Bryant, Arkansas
  - Study Site 220, Beverly Hills, California
  - Study Site 204, Fremont, California
  - Study Site 356, San Diego, California
  - Study Site 202, San Diego, California
  - Study Site 215, San Diego, California
  - Study Site 376, Santa Monica, California
  - Study Site 212, Clearwater, Florida
  - Study Site 210, Coral Gables, Florida
  - Study Site 331, Miami, Florida
  - Study Site 348, Miami, Florida
  - Study Site 222, North Miami Beach, Florida
  - Study Site 206, Sanford, Florida
  - Study Site 213, Boise, Idaho
  - Study Site 360, New Albany, Indiana
  - Study Site 207, South Bend, Indiana
  - Study Site 228, Louisville, Kentucky
  - Study Site 216, Louisville, Kentucky
  - Study Site 506, Ann Arbor, Michigan
  - Study Site 219, Clinton Township, Michigan
  - Study Site 209, Fridley, Minnesota
  - Study Site 371, Saint Joseph, Missouri
  - Study Site 227, Omaha, Nebraska
  - Study Site 201, East Windsor, New Jersey
  - Study Site 375, Forest Hills, New York
  - Study Site 500, New York, New York
  - Study Site 516, Bexley, Ohio
  - Study Site 211, Broomall, Pennsylvania
  - Study Site 345, Johnston, Rhode Island
  - Study Site 205, Murfreesboro, Tennessee
  - Study Site 182, College Station, Texas
  - Study Site 224, Houston, Texas
  - Study Site 359, Pflugerville, Texas
  - Study Site 339, Plano, Texas
  - Study Site 203, San Antonio, Texas
  - Study Site 223, Sugar Land, Texas
  - Study Site 226, Webster, Texas
  - Study Site 217, Norfolk, Virginia
  - Study Site 336, Richmond, Virginia

REFERENCES:
- [Derived] Pariser DM, Bagel J, Lebwohl M, Yosipovitch G, Chien E, Spellman MC. Serlopitant for psoriatic pruritus: A phase 2 randomized, double-blind, placebo-controlled clinical trial. J Am Acad Dermatol. 2020 Jun;82(6):1314-1320. doi: 10.1016/j.jaad.2020.01.056. Epub 2020 Jan 30. PMID 32007513

RESULTS

PARTICIPANT FLOW:
Groups:
- Serlopitant 5 mg: Subjects received a 3-tablet oral loading dose (15 mg) on the first day of the treatment period followed by a 5 mg dose of Serlopitant taken once daily by mouth for 8 weeks
- Placebo: Subjects received a 3-tablet oral loading dose on the first day of the treatment period followed by a Placebo tablet taken once daily by mouth for 8 weeks
Period: Overall Study
Arm/Group | Serlopitant 5 mg | Placebo
Started | 102 | 102
Completed | 88 | 90
Not Completed | 14 | 12
Not completed — Withdrawal by Subject | 10 | 6
Not completed — Lost to Follow-up | 4 | 5
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: The populations here represent the Full Analysis Set, not all randomized subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | Serlopitant 5 mg | Placebo | Total
Number analyzed (Participants) | 102 | 101 | 203
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.2 (15.2) | 46.7 (12.34) | 47.5 (13.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 62 | 110
  Male | 54 | 39 | 93
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29 | 31 | 60
  Not Hispanic or Latino | 73 | 70 | 143
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 3 | 4 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 12 | 6 | 18
  White | 84 | 89 | 173
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 102 | 101 | 203
WI-NRS [Mean (Standard Deviation); unit: units on a scale] — Worst Itch Numeric Rating Scale (WI-NRS). 11-point scale ranging from 0 (no itch) to 10 (worst itch imaginable). Higher scores indicate greater itch intensity. Subject-reported score from reflection on past 24 hours. The baseline was established by averaging 7 daily scores leading up to randomization.
  units on a scale | 8.303 (1.0277) | 8.082 (1.0588) | 8.193 (1.0466)

OUTCOME MEASURES:

1. Primary Outcome: WI-NRS 4-point Responder Rate at Week 8
Description: Worst Itch Numeric Rating Scale (WI-NRS). 11-point scale ranging from 0 (no itch) to 10 (worst itch imaginable). Higher scores indicate greater itch intensity. A 4-point responder is a subject who had at least a 4-point reduction in score between Baseline and Week 8.
Time Frame: 8 weeks
Population: These figures represent full analysis set.
Measure: Number; unit: % of subjects (incl. imputed data)
Arm/Group | Serlopitant 5 mg | Placebo
Number analyzed (Participants) | 102 | 101
% of subjects (incl. imputed data) | 33.29 | 21.07

2. Secondary Outcome: WI-NRS 4-point Responder Rate at Week 4
Description: Worst Itch Numeric Rating Scale (WI-NRS). 11-point scale ranging from 0 (no itch) to 10 (worst itch imaginable). Higher scores indicate greater itch intensity. A 4-point responder is a subject who had at least a 4-point reduction in score between Baseline and Week 4.
Time Frame: 4 weeks
Population: These figures represent full analysis set
Measure: Number; unit: percentage of subjects
Arm/Group | Serlopitant 5 mg | Placebo
Number analyzed (Participants) | 102 | 101
percentage of subjects | 20.78 | 11.49

3. Secondary Outcome: Change in WI-NRS From Baseline to Day 7
Description: Worst Itch Numeric Rating Scale (WI-NRS). 11-point scale ranging from 0 (no itch) to 10 (worst itch imaginable). Higher scores indicate greater itch intensity. The secondary outcome is the change in WI-NRS score at 7 days compared with Baseline.
Time Frame: Change from baseline to day 7
Population: These figures represent full analysis set
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Serlopitant 5 mg | Placebo
Number analyzed (Participants) | 102 | 101
units on a scale | -1.307 (1.8741) | -0.785 (1.8391)

4. Secondary Outcome: Change in WI-NRS From Baseline to Day 3
Description: Worst Itch Numeric Rating Scale (WI-NRS). 11-point scale ranging from 0 (no itch) to 10 (worst itch imaginable). Higher scores indicate greater itch intensity. The secondary outcome is the change in WI-NRS score at 3 days compared with Baseline.
Time Frame: 3 days
Population: These figures represent full analysis set.
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Serlopitant 5 mg | Placebo
Number analyzed (Participants) | 102 | 101
units on a scale | -0.702 (1.4111) | -0.461 (1.4060)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) and Serious Adverse Events (SAEs) were recorded from the first study drug administration through the Follow-up visit, for a total of approximately 10 weeks.
Description: The safety population is a subset of participants who received at least one dose of study medication with at least one post-baseline assessment or a reported treatment emergent adverse event. This population was analyzed based upon the actual treatment received.
Arm/Group | Serlopitant 5 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/102 | 1/100
Serious Adverse Events (participants affected / at risk) | 0/102 | 2/100
Other Adverse Events (participants affected / at risk) | 9/102 | 17/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Serlopitant 5 mg (N=102) | Placebo (N=100)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Serlopitant 5 mg (N=102) | Placebo (N=100)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 3 (4)
Nasopharyngitis (Infections and infestations) | 2 (2) | 6 (6)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 4 (4)
Headache (Nervous system disorders) | 3 (3) | 5 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-03-15): https://cdn.clinicaltrials.gov/large-docs/39/NCT03343639/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-09): https://cdn.clinicaltrials.gov/large-docs/39/NCT03343639/SAP_001.pdf